CLINICAL TRIAL: NCT03192813
Title: Safety and Efficacy Comparison Of Two TAVI Systems in a Prospective Randomized Evaluation II: A Randomized, Controlled, Non-inferiority Trial Evaluating Safety and Clinical Efficacy of the Symetis ACURATE Neo Compared to the Medtronic Evolut R Bioprosthesis in Transfemoral Transcatheter Aortic Valve Implantation
Brief Title: Safety and Efficacy Comparison Of Two TAVI Systems in a Prospective Randomized Evaluation II
Acronym: SCOPE II
Status: Completed | Type: Observational
Sponsor: Ceric Sàrl (Industry)
Collaborators: Symetis SA (Industry)
Responsible Party: Sponsor
Other Study IDs: SCOPE II
Record Dates: First submitted 2017-03-30; First posted 2017-06-20 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symetis ACURATE neo™ transfemoral TAVI system: Patient assigned to this group will be implanted with Symetis ACURATE neo™ transfemoral TAVI system.
  Interventions: Device: Symetis ACURATE neo™ transfemoral TAVI system
- Medtronic CoreValve Evolut R TAVI System: Patient assigned to this group will be implanted with Medtronic CoreValve Evolut R Transcatheter Aortic Valve Implantation (TAVI) System.
  Interventions: Device: Medtronic CoreValve Evolut R TAVI System

INTERVENTIONS:
Device: Symetis ACURATE neo™ transfemoral TAVI system — Symetis ACURATE neo™ transfemoral TAVI system: Support frame made of nitinol, supra-annular processed tri-leaflet porcine pericardial valve and an outer skirt to mitigate paravalvular regurgitation (manufactured by Symetis SA, Ecublens, Switzerland).
  Groups: Symetis ACURATE neo™ transfemoral TAVI system
Device: Medtronic CoreValve Evolut R TAVI System — Medtronic CoreValve Evolut R Transcatheter Aortic Valve Implantation (TAVI) System (or any future CE-marked Corevalve versions): The support frame is manufactured from nitinol, which has multilevel, self-expanding properties and is radiopaque. The bioprosthesis is manufactured by suturing valve leaflets and a skirt from porcine pericardium into a tri-leaflet configuration (manufactured by Medtronic CoreValve LLC, Santa Ana, USA).
  Groups: Medtronic CoreValve Evolut R TAVI System

SUMMARY:
Current care randomized clinical trial comparing the CE marked Symetis ACURATE neo™ Aortic Bioprosthesis and ACURATE TF™ Transfemoral Delivery System with the CE marked Medtronic CoreValve Evolut R TAVI system (or any future CE-marked CoreValve versions).

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVI) is an established and valuable treatment option for patients with severe symptomatic aortic stenosis and at high surgical risk for aortic valve replacement. The use of TAVI is rapidly expanding worldwide and its indications are widening into intermediate and lower risk populations. However, device comparisons by use of randomized trials are scarce in particular for newer generation transcatheter valves.

The Symetis ACURATE neo™, a self-expanding transcatheter valve delivered via transfemoral access, is a second-generation device that gained CE mark approval in June 2014.

The SCOPE-II trial will compare the safety and performance of the Symetis ACURATE neo™ with the self-expanding Medtronic Evolut R system, a widely used and well-established transcatheter heart valve, which obtained CE mark in 8NOV2006 and HAS approval on 13JAN2015.

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe symptomatic aortic stenosis defined by a mean aortic gradient > 40 mmHg or peak jet velocity > 4.0 m/s or an aortic valve area (AVA) < 1cm2 or AVA indexed to body surface area (BSA) of <0.6 cm2/m2
* Patient is symptomatic (heart failure with New York Heart Association (NYHA) Functional Class > I, angina or syncope)
* Patients are considered at high risk for mortality with conventional surgical aortic valve replacement as assessed by a Heart Team consisting of a cardiologist and surgeon or as confirmed by a logistic EuroSCORE I > 20% and / or STS score > 10%.
* Aortic annulus diameter ranging from 21 to 26mm and perimeter rage from 66 - 81.7mm , based on ECG-gated multi-slice computed tomographic measurements. Findings of TTE, TEE and conventional aortography should be integrated in the anatomic assessment.
* Arterial aorto-iliac-femoral axis suitable for transfemoral access as assessed by conventional angiography and/or multi-detector computed tomographic angiography (access vessel diameter ≥ 6mm)
* Patient understands the purpose, the potential risks as well as benefits of the trial and is willing to participate in all parts of the follow-up
* Patient age 75 years or older
* Patient has given written consent to participate in the trial

Exclusion Criteria:

* Severely reduced left ventricular (LV) function (ejection fraction <20%)
* Pre-existing prosthetic heart valve in aortic and/or mitral position
* Participation in another trial, which would lead to deviations in the preparation or performance of the intervention or the post-implantation management from this protocol
* Severe coagulation conditions
* Inability to tolerate anticoagulation therapy
* Contraindication to contrast media or allergy to nitinol
* Active infection, including endocarditis
* Congenital aortic stenosis or unicuspid or bicuspid aortic valve
* Non-valvular aortic stenosis
* Hypertrophic obstructive cardiomyopathy
* New or untreated echocardiographic evidence of intracardiac mass, thrombus, or vegetation
* Non-calcific acquired aortic stenosis
* Severe eccentricity of calcification
* Anatomy not appropriate for transfemoral implant due to size, disease and degree of calcification or tortuosity of the aorta or ilio-femoral arteries
* Severe mitral regurgitation

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 764 patients presenting with severe symptomatic aortic stenosis with the indication for TAVI, as agreed by the Heart Team. If all eligibility criteria and none of the exclusion criteria are fulfilled, patients will be allocated in a 1:1 ratio to either the Symetis ACURATE neo™ or the Medtronic CoreValve Evolut R (or any future CE-marked CoreValve versions) by permuted block randomization.
Sampling Method: Probability Sample
Enrollment: 796 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality or stroke rates | 1 year
  The primary objective is to compare the composite of all-cause mortality or stroke rates at 1 year (powered for non-inferiority).

SECONDARY OUTCOMES:
New permanent pacemaker rate | 30 days
  The first secondary objective is to compare the new permanent pacemaker rate at 30 days (powered for superiority).
All cause mortality at 30 days | 30 days
  All cause mortality
Stroke at 30 days | 30 days
  Stroke
Valve malpositioning at 30 days | 30 days
  Valve malpositioning
Peri-procedural myocardial infarction at 30 days | 30 days
  Peri-procedural myocardial infarction
Cardiac Tamponade at 30 days | 30 days
  Cardiac Tamponade
Implantation of multiple valves (TAV-in-TAV deployment) at 30 days | 30 days
  Implantation of multiple valves (TAV-in-TAV deployment)
Annular rupture/dissection at 30 days | 30 days
  - Annular rupture/dissection
Left ventricular perforation at 30 days | 30 days
  - Left ventricular perforation
Conversion to open heart surgery at 30 days | 30 days
  - Conversion to open heart surgery
Intra-procedural mortality (during index procedure) | Procedurally
  - Intra-procedural mortality (during index procedure)
Procedural mortality (up to 72 hours after procedure) | Procedurally and up to 72 hours post-procedurally
  - Procedural mortality (up to 72 hours after procedure)
Mortality (cardiac/non-cardiac) at 30 days and 1 year | 30 days and 1 year
  - Mortality (cardiac/non-cardiac)
All stroke (disabling/non disabling) at 30 days and 1 year | 30 days and 1 year
  - All stroke (disabling/non disabling)
Composite of all-cause mortality or disabling stroke at 30 days and 1 year | 30 days and 1 year
  - Composite of all-cause mortality or disabling stroke
Hospitalization for valve-related symptoms or worsened congestive heart at 30 days and 1 year | 30 days and 1 year
  - Hospitalization for valve-related symptoms or worsened congestive heart failure
Life-threatening/major bleeding at 30 days and 1 year | 30 days and 1 year
  - Life-threatening/major bleeding (BARC 3b or more)
Myocardial infarction at 30 days and 1 year | 30 days and 1 year
  - Myocardial infarction
Valve related dysfunction requiring repeat procedure at 30 days and 1 year | 30 days and 1 year
  - Valve related dysfunction requiring repeat procedure (BAV, TAVI or SAVR)
Endocarditis at 30 days and 1 year | 30 days and 1 year
  - Endocarditis
Valve thrombosis at 30 days and 1 year | 30 days and 1 year
  - Valve thrombosis
New AV-conduction disturbances at 30 days and 1 year | 30 days and 1 year
  - New AV-conduction disturbances (LBBB only)
New pacemaker implantation at 1 year | 1 year
  - New pacemaker implantation at 1 year
Any arrhythmia resulting in hemodynamic instability or requiring therapy at 30 days and 1 year | 30 days and 1 year
  Any arrhythmia resulting in hemodynamic instability or requiring therapy
VARC-2 combined endpoints at 30 days | 30 days
  Composite of device success, early safety, clinical efficacy and time-related valve safety
Time-related valve safety at 1 year | 1 year
  Time-related valve safety
Echocardiographic endpoint (1) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - Structural valve deterioration
Echocardiographic endpoint (2) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - Prosthetic aortic valve stenosis
Echocardiographic endpoint (3) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - Patient prosthesis mismatch
Echocardiographic endpoint (4) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - Aortic regurgitation (grading), proportion of more than mild regurgitation
Echocardiographic endpoint (5) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - Intended valve performance: No prosthesis mismatch, mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, without moderate or severe prosthetic valve aortic regurgitation.
Echocardiographic endpoint (6) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - Systolic LV ejection fraction
Echocardiographic endpoint (7) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - LV diastolic function
Echocardiographic endpoint (8) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - Left atrial volume
Echocardiographic endpoint (9) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - Right ventricular (RV) dimension and function
Echocardiographic endpoint (10) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - Right atrial (RA) area
Echocardiographic endpoint (11) | Post-procedurally [day 1 to 7], at 30 days, 1 year
  - RV/RA-ratio and estimated systolic pulmonary arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tamburino, Prof, MD, PhD, Principal Investigator — Cardiology Division and Cardio-Thoracic & Vascular Department, Ferrarotto & Policlinico Hospitals, University of Catania, Italy; Sabine Bleiziffer, MD, Principal Investigator — Herz- und Diabeteszentrum NRW, Bad Oeynhausen, Germany
Locations (23):
- Heart Center, Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- France (4):
  - CHRU Brest Cavale Blanche, Brest
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hôpital Jacques Cartier, Massy
  - Clinique Pasteur, Toulouse
- Germany (11):
  - University Hospital Aachen, Aachen
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Herzzentrum Brandenburg, Immanuel Klinikum Bernau, Bernau bei Berlin
  - St.-Johannes-Hospital, Dortmund
  - Technische Universität Dresden, Dresden
  - Elisabeth-Krankenhaus Essen, Essen
  - Goethe-University Frankfurt, Frankfurt
  - Herzzentrum Leipzig - Universitätsklinik, Leipzig
  - Deutsches Herzzentrum München des Freistaates Bayern, Munich
  - Klinik für Herz- & Kreislauferkrankungen - Deutsches Herzzentrum München, Munich
- Italy (4):
  - University of Catania, Ferrarotto Hospital, Catania
  - Istituto Clinico Humanitas, Rozzano- (MI)
  - IRCCS Policlinico San Donato, San Donato
  - Ospedale San Raffaele, San Raffaele
- Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, Spain
- United Kingdom (2):
  - Brighton and sussex University hospital NHS trust, Brighton, England
  - The Leeds Teaching Hospitals NHS TRUST, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tamburino C, Bleiziffer S, Thiele H, Scholtz S, Hildick-Smith D, Cunnington M, Wolf A, Barbanti M, Tchetche D, Garot P, Pagnotta P, Gilard M, Bedogni F, Van Belle E, Vasa-Nicotera M, Chieffo A, Deutsch O, Kempfert J, Sondergaard L, Butter C, Trillo-Nouche R, Lotfi S, Mollmann H, Joner M, Abdel-Wahab M, Bogaerts K, Hengstenberg C, Capodanno D. Comparison of Self-Expanding Bioprostheses for Transcatheter Aortic Valve Replacement in Patients With Symptomatic Severe Aortic Stenosis: SCOPE 2 Randomized Clinical Trial. Circulation. 2020 Dec 22;142(25):2431-2442. doi: 10.1161/CIRCULATIONAHA.120.051547. Epub 2020 Oct 15. PMID 33054367